CLINICAL TRIAL: NCT01069068
Title: Assessment of the Impact of a Stepped Mouthpiece on the Upper Airways Measured Through Acoustic Pharyngometry
Status: Completed | Type: Observational
Sponsor: Doctor's Directive Strategies Inc. (Other)
Responsible Party: Principal Investigator, Dr John Viviano, Principal Investigator, Doctor's Directive Strategies Inc.
Other Study IDs: RDD-2009-001
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: To evaluate the effect of advancing Jaw on airway dimension
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Mandibular advancements during tidal breathing, achieved through a stepped mouthpiece design, affect the size of the upper airways in subjects with and without Obstructive Sleep Apnea.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent to participate in the study.
* Adult male or female subjects over 18 years of age who have or have not been diagnosed with OSA.
* Subjects claiming no history of OSA should take the Epworth questionnaire and obtain a result less than 10.
* Subjects must satisfy the study investigator about their fitness to participate in the study.
* Subjects must be available to complete the study.

Exclusion Criteria:

* Subjects not compliant with the instructions for use of the stepped mouthpiece and the study procedures.
* Subjects who have participated in a clinical trial in the previous month.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be performed as an open investigation including 60 subjects. The 60 subjects will be stratified such that 30 subjects should have been diagnosed with OSA, and 30 subjects should not have been diagnosed with OSA.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To measure the impact of different horizontal mandibular advancements, achieved through a stepped mouthpiece design, on the size of the upper airways in subjects with and without Obstructive Sleep Apnea (OSA). | one 60 minute session

SECONDARY OUTCOMES:
Assessment of the habitual mandibular position in (edge-to-edge, millimetres) relation to the front upper teeth | one 60 minute session
Measurement of the upper airways through acoustic pharyngometry during slow and deep breathing while the subject uses a stepped mouthpiece. The acoustic pharyngometry measurement will be performed at mid inhalation | one 60 minute session
Assessment of the most comfortable position when using the stepped mouthpiece during both "tidal" and "slow and deep breathing". The scoring of the "comfortable position" will be performed through a Likert-style questionnaire | one 60 minute session
The most "comfortable position" established as outlined above will be evaluated for comfort while holding that position for 3 minutes. After the 3 minutes, the subject's level of comfort will be re-evaluated through a Likert-style questionnaire | one 60 minute session

CONTACTS AND LOCATIONS:
Overall Officials: John S Viviano, DDS, Principal Investigator — Dr John Viviano
Locations (1):
- Dr John Viviano and Associates, Mississauga, Ontario, Canada